CLINICAL TRIAL: NCT04013724
Title: Efficacy of a Group Tobacco Cessation Behavioral Intervention Among Tobacco Users With Concomitant Mental Illness in Kenya: Protocol for a Controlled Clinical Trial
Brief Title: Efficacy of Group Tobacco Cessation Interventions Among Tobacco Users With Mental Illness: Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nairobi (Other)
Responsible Party: Principal Investigator, Yvonne Olando, Clinical Psychologist, University of Nairobi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P641/09/2016
Record Dates: First submitted 2019-07-02; First posted 2019-07-10 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Mental Illness
Keywords: Tobacco cessation, mental illness, tobacco dependence, Kenya
MeSH Terms: conditions — Mental Disorders; Tobacco Use Cessation; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: The participants in the intervention group were introduced to a structured group tobacco cessation program. They met twice a month, for a period of 3 months, then were followed up once a month for a period of 3 months. Each meeting session lasted for a period of 45 minutes. They shared their feelings, and experiences with cessation attempt at the beginning of each session. The facilitator then documented their quit attempts, any changes in numbers of cigarettes smoked, and any challenges with cessation attempts noted. The facilitator then introduced the topic of the day and facilitated discussion on the same. Where skills practice was involved, the facilitator demonstrated to the participants how to apply the skill.
Who Masked: Outcomes Assessor
Masking Description: At the group assessments (Weeks 4, 12, and 26), participants who reported continued tobacco use abstinence and consented to a saliva test were tested using a nicotine cotinine strip (Devon Medical: Nicotine/tobacco test kit). The saliva tests were evaluated by the nurses working at the hospital who were blinded to treatment allocation and were not otherwise part of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The behavioral group intervention consisted of 6 sessions over 12 weeks and were led by 2 trained facilitators, followed by monthly group meetings from weeks 14 to 26. This program was adapted from the Royal Australian College of General Practitioners' Supporting Smoking Cessation Guide for Health Professionals17 and the World Health Organization's Strengthening Health Systems for Treating Tobacco Dependence in Primary Care training package.18
  The topics that were explored during the group sessions include:
  1. Introduction to the Program and Reasons to Quit
  2. Benefits of Quitting and Understanding Why We Smoke and Ways of Quitting
  3. Withdrawal Symptoms and Social Support
  4. Dealing with Stress and Anxiety and Coping with Depression
  5. Assertiveness Training and Anger Management
  6. Tobacco-Free Lifestyle and Dealing with High Risk Situations
  Interventions: Behavioral: Group tobacco cessation interventions
- Control (No Intervention): The control group was provided questionnaires to fill at the end of Weeks 4, 12, and 26. During the rest of the study, they continued receiving usual care, including clinical care at CSAT.

INTERVENTIONS:
Behavioral: Group tobacco cessation interventions — Group Session Week 1 Participants were introduced to the specific components of the group behavioral intervention. Participants shared their expectations and experiences in their goal of tobacco cessation.
  Group Sessions Weeks 2-11 Participants set their anticipated quit date on the 2nd week. During weeks 2 through 11, before the start of the session, feelings of participants were explored, the previous week's self-reported tobacco consumption or cessation attempt was recorded. The topic of each week was explored first by lecture to explain the topic, and then group members took turns sharing their experiences on the topic.
  Group Sessions Weeks 14-26 Behavioral group sessions weeks 14-26 were conducted once a month. Each session began with a round of discussion on how participants were feeling about their cessation attempts, including any challenges they had experienced. The self-reported amount of tobacco used and quit attempts were documented.
  Arms: Intervention group

SUMMARY:
The study seeks to provide group tobacco cessation interventions among patients who use tobacco, and who attend Mathari National referral hospital on outpatient follow up. They will also be assessed on changes in quality of life before and after provision of the intervention.

DETAILED DESCRIPTION:
All patients who walked in for follow-up after hospital discharge for a primary mental health diagnosis were informed of the study and were invited to participate. Informed consent was obtained from individuals who had capacity to provide informed consent in the presence of the clinicians working with the participants to ensure they understood the study requirements. Individuals who did not have capacity to provide informed consent were not recruited to minimize potential risks to this vulnerable population. After providing informed consent, participants were asked to complete the Fagerstrom tobacco use test. Participants were then asked to complete sociodemographic questionnaire and the World Health Organization (WHO) quality of life questionnaire. This screening and recruitment continued until the number of participants who provided informed consent reached 100.

Randomization/Allocation Participants were recruited in clusters of 10 for allocation into the intervention and control groups. The first 10 participants formed group 1, and the next 10 participants formed group 2. Group 1 became the first intervention group, while group 2 became the first control group. This procedure continued until all 10 groups were formed (5 intervention and 5 control groups).

Participants were followed up clinically for ongoing mental health care on their regular clinic days.

Study intervention 5As-based brief advice was offered to the intervention group participants by the study team who were trained by YO. This brief advice consisted of an individual session lasting approximately 5 minutes for each participant immediately after their consent had been obtained. The focus of the 5As was to enable the therapist know the immediate concern of each participant and to enable adequate support when the particular issues were raised during the group intervention sessions. The behavioral group intervention consisted of 6 sessions over 12 weeks and were led by 2 trained facilitators, followed by monthly group meetings from weeks 14 to 26. This program was adapted from the Royal Australian College of General Practitioners' Supporting Smoking Cessation Guide for Health Professionals17 and the World Health Organization's Strengthening Health Systems for Treating Tobacco Dependence in Primary Care training package.18

The topics that were explored during the group sessions include:

1. Introduction to the Program and Reasons to Quit
2. Benefits of Quitting and Understanding Why We Smoke and Ways of Quitting
3. Withdrawal Symptoms and Social Support
4. Dealing with Stress and Anxiety and Coping with Depression
5. Assertiveness Training and Anger Management
6. Tobacco-Free Lifestyle and Dealing with High Risk Situations

Group Session 1 (Week 1) On the first session, participants were introduced to the study program and specific components of the group behavioral intervention. Participants shared their expectations and experiences in their goal of tobacco cessation. The estimated time for group session 1 was 30-45 minutes.

Group Sessions 2-6 (Weeks 2-11) Participants set their anticipated quit date on the 2nd week, which was their second session. During weeks 2 through 11, before the start of the session, feelings of participants were explored, the previous week's self-reported tobacco consumption or cessation attempt was recorded. The topic of each week was explored first by lecture to explain the topic, and then group members took turns sharing their experiences on the topic.

Group Sessions 7-9 (Weeks 14-26) Participants continued attending the CSAT outpatient and ward follow-up programs during this period. Behavioral group sessions 7-9 (weeks 14-26) were conducted once a month by the facilitators whereby each session was begun with a round of discussion on how participants were feeling about their cessation attempts, including any challenges they had experienced. The self-reported amount of tobacco used and quit attempts were documented. The study team also documented the challenges raised and tried to offer practical and supportive therapy for the challenges.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and above.
2. History of tobacco use for more than 6 months.
3. A Fagerstrom score of 6 and above, which is a threshold consistent with dependence.16
4. Currently on outpatient follow up treatment for a diagnosed mental health condition.
5. Willing to be part of the study for 6 months.

Exclusion Criteria:

1. Patients on nicotine replacement therapy (NRT) or other pharmacotherapy for tobacco cessation.
2. Patients currently experiencing severe psychotic episodes judged by their treating health care provider.
3. Patients who would not be able to commit to the group sessions, defined as those who would not be able to attend group sessions for any reason, including transport-related reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Self reported continued tobacco use abstinence | Week 4, 12 and 26
  The study's primary outcome was self-reported continuous tobacco use abstinence, biochemically verified.
Health related quality of life | Week 26
  Secondary outcome assessed included changes in health related quality of life as assessed by WHOQOL

SECONDARY OUTCOMES:
Quit attempts | Week 4, 12 and 26
  Secondary outcomes assessed included self reported quit attempts
Reduction in amounts used | Week 4, 12 and 26
  Secondary outcome assessed included change in amount of cigarettes smoked or tobacco used, as reported by participants

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Olando, Principal Investigator — University of Nairobi
Locations (1):
- Mathari Treatment and Referral Hospital, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data sharing may be considered upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after analysis is complete. This should be in November 2019.
Access Criteria: On request

REFERENCES:
- [Background] World Health Organization. International Classification of Diseases (ICD-10) and Health Problems. Geneva, Switzerland. 2015
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders (Fifth version). Arlington, VA: American Psychiatric Association. 2013
- [Background] Action on Smoking and Health (ASH) Fact sheet. Smoking and Mental Health. 2016. Available at: http://ash.org.uk/category/information-and-resources/fact-sheets/. Accessed 15 May 2019.
- [Background] Heiligenstein E, Smith SS. Smoking and mental health problems in treatment-seeking university students. Nicotine Tob Res. 2006 Aug;8(4):519-23. doi: 10.1080/14622200600789718. PMID 16920649
- [Background] Brown C. Tobacco and Mental Health: A review of the literature. Edinburgh: ASH Scotland. 2004
- [Background] Royal College of Psychiatrists. Liaison Psychiatry for acute hospital: Integrated mental and physical healthcare. London: College Report, Royal College of Psychiatrists. 2013
- [Background] John U, Meyer C, Rumpf HJ, Hapke U. Smoking, nicotine dependence and psychiatric comorbidity--a population-based study including smoking cessation after three years. Drug Alcohol Depend. 2004 Dec 7;76(3):287-95. doi: 10.1016/j.drugalcdep.2004.06.004. PMID 15561479
- [Background] Weir, K. Smoking and mental illness. American Psychological Association Science Watch. 2013; 44 (6): 36.
- [Background] Hall SM, Prochaska JJ. Treatment of smokers with co-occurring disorders: emphasis on integration in mental health and addiction treatment settings. Annu Rev Clin Psychol. 2009;5:409-31. doi: 10.1146/annurev.clinpsy.032408.153614. PMID 19327035
- [Background] Cavazos-Rehg PA, Breslau N, Hatsukami D, Krauss MJ, Spitznagel EL, Grucza RA, Salyer P, Hartz SM, Bierut LJ. Smoking cessation is associated with lower rates of mood/anxiety and alcohol use disorders. Psychol Med. 2014 Sep;44(12):2523-35. doi: 10.1017/S0033291713003206. PMID 25055171
- [Background] Prochaska JJ, Delucchi K, Hall SM. A meta-analysis of smoking cessation interventions with individuals in substance abuse treatment or recovery. J Consult Clin Psychol. 2004 Dec;72(6):1144-56. doi: 10.1037/0022-006X.72.6.1144. PMID 15612860
- [Background] Gulliver SB, Wolfsdorf BA, Morissette SB. Treating tobacco dependence: Development of a smoking cessation treatment program for outpatient mental health clinics. Cogn Behav Pract. 2004; 11, 315-330
- [Background] Morris CD, Tedeschi GJ, Waxmonsky JA, May M, Giese AA. Tobacco quitlines and persons with mental illnesses: perspective, practice, and direction. J Am Psychiatr Nurses Assoc. 2009 Feb;15(1):32-40. doi: 10.1177/1078390308330050. PMID 21665792
- [Background] Tsoi DT, Porwal M, Webster AC. Interventions for smoking cessation and reduction in individuals with schizophrenia. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD007253. doi: 10.1002/14651858.CD007253.pub3. PMID 23450574
- [Background] Bron C, Zullino D, Besson J, Borgeat F. [Smoking in psychiatry, a neglected problem]. Praxis (Bern 1994). 2000 Oct 19;89(42):1695-9. French. PMID 11105610
- [Background] Fagerstrom KO, Schneider NG. Measuring nicotine dependence: a review of the Fagerstrom Tolerance Questionnaire. J Behav Med. 1989 Apr;12(2):159-82. doi: 10.1007/BF00846549. PMID 2668531
- [Background] The Royal Australian College of General Practitioners. Supporting smoking cessation: Guide for health professionals. Royal College of General Practitioners. Melbourne, Australia. 2011
- [Background] World Health Organization. Strengthening health systems for treating tobacco dependence in primary care: Building capacity for tobacco control: Training package.Geneva, Switzerland. 2013
- [Background] Bentz CJ, Bayley KB, Bonin KE, Fleming L, Hollis JF, Hunt JS, LeBlanc B, McAfee T, Payne N, Siemienczuk J. Provider feedback to improve 5A's tobacco cessation in primary care: a cluster randomized clinical trial. Nicotine Tob Res. 2007 Mar;9(3):341-9. doi: 10.1080/14622200701188828. PMID 17365766
- [Background] Buckley TC, Mozley SL, Holohan DR, Walsh K, Beckham JC, Kassel JD. A psychometric evaluation of the Fagerstrom Test for Nicotine Dependence in PTSD smokers. Addict Behav. 2005 Jun;30(5):1029-33. doi: 10.1016/j.addbeh.2004.09.005. PMID 15893100
- [Background] Study protocol for the World Health Organization project to develop a Quality of Life assessment instrument (WHOQOL). Qual Life Res. 1993 Apr;2(2):153-9. PMID 8518769
- [Background] Mas-Exposito L, Amador-Campos JA, Gomez-Benito J, Lalucat-Jo L; Research Group on Severe Mental Disorder. The World Health Organization Quality of Life Scale Brief Version: a validation study in patients with schizophrenia. Qual Life Res. 2011 Sep;20(7):1079-89. doi: 10.1007/s11136-011-9847-1. Epub 2011 Feb 3. PMID 21290191
- [Derived] Olando Y, Kuria M, Mathai M, Huffman MD. Efficacy of a group tobacco cessation behavioral intervention among tobacco users with concomitant mental illness in Kenya: protocol for a controlled clinical trial. BMC Public Health. 2019 Dec 18;19(1):1700. doi: 10.1186/s12889-019-8040-2. PMID 31852536